CLINICAL TRIAL: NCT00781716
Title: Comparison of Safety and Efficacy of CYPHER® Sirolimus Stent and ENDEAVOR® Zotarolimus Stent in Patients With Acute ST Elevation Myocardial Infarction and Analysis of Current Status of Emergency PCI Green Channel for Patients With ST Elevation Myocardial Infarction in China
Brief Title: Safety and Efficacy Study of CYPHER® Sirolimus Stent and ENDEAVOR® Zotarolimus Stent in Patients With Acute ST Elevation Myocardial Infarction (STEMI) and Analysis of Current Status of Emergency PCI Green Channel for STEMI Patients in China
Acronym: CREST-MI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Dr. LeFeng Wang/Director of the Cath Lab, Beijing Chao Yang Hospital Heart Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Version 1.0-Sep 10, 2008
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Myocardial Infarction; Coronary Artery Disease
Keywords: ST elevation myocardial infarction; Drug eluting stents
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease; ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cypher Stent (Active Comparator): Cypher Sirolimus-Eluting Coronary Stent System
  Interventions: Device: Drug eluting coronary stent system
- Endeavor Stent (Active Comparator): Endeavor Zotarolimus-Eluting Coronary Stent System
  Interventions: Device: Drug eluting coronary stent system

INTERVENTIONS:
Device: Drug eluting coronary stent system — Cypher Sirolimus-Eluting Coronary Stent System vs Endeavor Zotarolimus-Eluting Coronary Stent System

SUMMARY:
This study is to compare the clinical effect of CYPHER® stent and ENDEAVOR® stent in patients with acute ST elevation myocardial infarction. It also aims to analyze the current status of emergency PCI green channel (time taken from door→ hospital→ PIC sign-off→ needle→ balloon) for patients with ST elevation myocardial infarction in China.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be ≥18 years and ≤75 of age.
2. Prolonged, continuous (≥ 30 min) chest pain despite nitrate and: (1) ST-segment elevation ≥ at least 2 leads, with reciprocal ST-segment elevation ≥ 0.05mv and precordial leads ST-segment elevation ≥ 0.01mv, or (2) newly developed left bundle branch block
3. Symptoms ≥ 30 min and ≤12 hours
4. The patient has consented to participate and has authorized the collection and release of his medical information by signing the "Patient Informed Consent Form"
5. All lesions requiring interventions in one or more native coronary arteries are amendable for implantation of one or more Cypher® Sirolimus-Eluting Coronary Stent System or Endeavor® Zotarolimus-Eluting Coronary Stent
6. The patient or guardian is willing and able to cooperate with study procedures and required follow up visits.

Exclusion Criteria:

1. Pregnant and breast-feeding female and female of childbearing potential, who possibly plan to become pregnant any time after enrollment into this study.
2. Systemic (intravenous) Sirolimus use within 12 months.
3. Patients with hypersensitivity or allergies to one of the drugs or components indicated in the Instructions for Use of either stents.
4. History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or will refuse blood transfusions.
5. Gastrointestinal or genitourinary bleeding within the prior 3 months, or major surgery within 2 months.
6. Current platelet count <100 x 10^9cells/L or Hgb <10 g/dL.
7. Fibrinolytic therapy for current MI treatment
8. Previous coronary intervention on target vessel or post-CABG vessel disease
9. Transplant patients
10. Patients with EF<25%
11. Patients with cardiogenic shock; with a life expectancy shorter than 12 months
12. Severe kidney dysfunction: Creatinine level ≥2.0mg/dL or dependence on dialysis.
13. Severe hepatic dysfunction (AST and ALT ≥ 3 times upper normal reference values).
14. The patient is currently, and during the CREST-MI Study, participating in another investigational device or drug study that clinically interferes with the CREST-MI study endpoints; or requires coronary angiography or other coronary artery imaging procedures. The patient may only be enrolled in the CREST-MI Study once.
15. Severe tortuous or calcified vessel; stent can not or has difficulty to go through; blood vessel diameter is smaller than the minimum stent diameter available; patients unsuitable for stent implantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1020 (Estimated)
Dates: Start 2008-10; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events defined as death, MI (Q wave and non-Q wave), emergent cardiac bypass surgery, or target lesion revascularization (repeat PTCA or CABG) | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: LeFeng Wang, MD, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chaoyang Hospital Heart Center, Beijing, BJ, China